CLINICAL TRIAL: NCT05806918
Title: A Multicenter, Randomized, Double-blind, Controlled, Non-inferiority Phase III Clinical Trial of Recombinant Human Interferon Alpha-2b Gel (ZK-A03) in Treatment of Herpes Zoster Before and After the Alteration of the Active Ingredient Manufacturer
Brief Title: Non-inferiority Study of ZK-A03 in Treatment of Herpes Zoster Before and After the Alteration of the Active Ingredient Manufacturer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZK-A03-LEES-2023-01
Record Dates: First submitted 2023-03-20; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Interferon α-2b Gel (After the Alteration) (Experimental)
  Interventions: Drug: Recombinant Human Interferon α-2b Gel (After the Alteration)
- Recombinant Human Interferon α-2b Gel (Before the Alteration) (Active Comparator)
  Interventions: Drug: Recombinant Human Interferon α-2b Gel (Before the Alteration)

INTERVENTIONS:
Drug: Recombinant Human Interferon α-2b Gel (After the Alteration) — Recombinant human interferon α-2b gel (after the alteration of the active ingredient manufacturer) will be applied to the lesions as a thin layer, at the frequency of four times a day, together with the therapy of valaciclovir hydrochloride.
  Arms: Recombinant Human Interferon α-2b Gel (After the Alteration)
Drug: Recombinant Human Interferon α-2b Gel (Before the Alteration) — Recombinant human interferon α-2b gel (before the alteration of the active ingredient manufacturer) will be applied to the lesions as a thin layer, at the frequency of four times a day, together with the therapy of valaciclovir hydrochloride.
  Arms: Recombinant Human Interferon α-2b Gel (Before the Alteration)

SUMMARY:
The goal of this clinical trail is to demonstrate the non-inferiority of recombinant human interferon α-2b gel (ZK-A03) after changing the manufacturer of the active ingredient in patients with herpes zoster.

This double-blind study will enroll approximately 368 adult patients with herpes zoster in China. Eligible patients will be assigned randomly at a 1:1 ratio.

For each patient who is included, treatment may last up to 10 days. During the study, subjects will be treated with recombinant human interferon α-2b gel (either before or after the alteration of the active ingredient manufacturer), at a frequency of four times a day, together with a background therapy of valaciclovir hydrochloride.

ELIGIBILITY:
Main Inclusion Criteria:

1. Men and women aged between 18 and 70 years old.
2. Diagnosed as herpes zoster.
3. Time to appearance of lesions ≤ 72 hours prior to the first dosing (lesions may represent as: erythema, papules or blisters), lesion area ≤ 3% body surface area (BSA).
4. Self-rated Numerical Rating Scale (NRS) in pain ≤ 6.
5. Negative serum pregnancy test for women of reproductive age. Birth control from first dosing until 1 month after last dosing for all men and women of reproductive age.
6. Subjects must have signed an informed consent form (ICF).

Main Exclusion Criteria:

1. Diagnosed as herpes zoster on face, visceral herpes zoster, herpes zoster meningitis, disseminated herpes zoster, zoster sine herpete or blood blisters and necrosis.
2. The lesion is complicated with other skin diseases that may affect the evaluation of efficacy,
3. Skin lesions combined with severe bacterial or fungal infections.
4. Use of antiviral or analgesic therapy for herpes zoster within 2 weeks prior to the first dosing.
5. Known allergies to recombinant human interferon α-2b and chemical structure analogs, valaciclovir or history of any drug, food or other allergy.
6. Liver and/or renal disfunction，ie. Alanine aminotransferase (ALT), Aspartate transaminase (AST) > 2 times of upper normal limit（ULN）; Creatinine Clearance Rate (CCR) < 50 L/min.
7. Combined with immunodeficiency disease or require long-term glucocorticoid or immunosuppressive drugs.
8. Combined with severe cardiovascular, respiratory, gastrointestinal or neurological disorders and remains unstable after treatment.
9. History of psychiatric illness or inability to fully comply to the protocol.
10. Use of another investigational product within 4 weeks prior to the first dosing.
11. Pregnant or lactating women.
12. Other conditions deemed by the investigator to be inappropriate for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate at visit 4 (Day 7) | 7 Days
  Clinical cure is defined as all blisters being dry and crustosus without erosion or ulceration.

SECONDARY OUTCOMES:
Clinical cure rate at visit 3 (Day 4), and visit 5 (Day 11) | 11 Days
  Clinical cure is defined as all blisters being dry and crustosus without erosion or ulceration.
Time to which new blisters stop appearing | 11 Days
  The time from the first day of medication (D1) to the cessation of new blisters.
The time to beginning of crusting. | 11 Days
  The time from the first day of medication (D1) to the beginning of crusting.
The time to which all blisters are crustosus. | 11 Days
  The time from the first day of medication (D1) to the crustosus of all blisters.
The pain improvement rate at visit 4 (Day 7) | 7 Days
  Pain change of ≥1 from baseline is considered as pain improvement.

IPD SHARING:
Plan to Share IPD: No